CLINICAL TRIAL: NCT05516329
Title: A Study to Assess the Diagnostic Performance of 18F-Thretide PET/CT in Men With Prostate Cancer
Brief Title: Study of 18F-Thretide PET/CT in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director of Nuclear Medicine Department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-PSMA
Record Dates: First submitted 2022-08-04; First posted 2022-08-25 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Thretide Injection (Experimental): 7±1 mCi (259±37 MBq) IV injection of 18F-Thretide
  Interventions: Drug: A single dose of 7±1 mCi (259±37 MBq) IV injection of 18F-Thretide

INTERVENTIONS:
Drug: A single dose of 7±1 mCi (259±37 MBq) IV injection of 18F-Thretide — The patients will be intravenously injected with 18F-Thretide and undergo PET/CT scan at 60~120 min after the injection.

SUMMARY:
This study evaluates the diagnostic performance and safety of 18F-Thretide PET/CT in patients with biopsy proven prostate cancer who has no any form of therapy against prostate caner or suspected recurrence of prostate cancer who have negative or equivocal findings on conventional imaging.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) is overexpressed in most cases of prostate cancer and is potentially associated with metastasis and progression of prostate cancer. Compared with 68Ga, the PET radionuclide 18F exhibits several advantages. 18F-Thretide (18F-labeled PSMA ligand) has been studied for preclinical evaluation and Pilot Clinical Study. This study evaluates the diagnostic performance and safety of 18F-Thretide PET/CT in patients with with biopsy proven prostate cancer who has no any form of therapy against prostate caner or suspected recurrence of prostate cancer who have negative or equivocal findings on conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age;
* For patients with newly diagnosed prostate cancer : (1) adult patients with PCa confirmed by biopsy; (2) no any form of therapy against PCa within last three months; (3) planned surgical treatment;
* For patients with suspected recurrence of prostate cancer: (1)Histopathologically confirmed prostate adenocarcinoma per original diagnosis, with subsequent definitive therapy; (2)Suspected recurrence of prostate cancer based on rising PSA after definitive therapy on the basis of: Post-radical prostatectomy: Detectable or rising PSA level ≥ 0.2 ng/mL with a confirmatory PSA ≥ 0.2 ng/mL ; or Post-radiation therapy, cryotherapy, or brachytherapy: Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir;
* Life expectancy ≥3 months as determined by the investigator;
* Able and willing to provide informed consent and comply with protocol requirements.

Exclusion Criteria:

* Known allergic history to fluoride 18F-Thretide injection and/or 99mTc-MDP or its excipients;
* Patients who cannot tolerate intravenous administration (such as a history of needle sickness or blood sickness);
* Those who are not suitable for or unable to complete PET or other imaging examinations due to special reasons, including claustrophobia and radiophobia, etc.
* Practitioners requiring prolonged exposure to radioactive conditions;
* Serious diseases of the heart, kidney, lung, vascular, nervous and psychiatric systems, immune deficiency diseases and hepatitis/cirrhosis;
* Have been diagnosed with clinical recurrence of prostate cancer;
* Patients receiving ADT treatment or chemotherapy;
* Patients who participated in clinical trials of radiopharmaceuticals within the previous 1 year;
* Participated in other interventional clinical trials within 1 month prior to screening;
* There are other conditions that the researcher considers inappropriate to participate in this study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
detection rate at the patient level | Within 60 days following 18F-Thretide PET/CT
  The Difference in detection rate of 18F-Thretide PET/CT at the patient level compared with MRI, CT, or bone scanning. Within 60 days following 18F-Thretide PET/CT imaging, either MRI, CT, or bone scanning will be performed.
detection rate at the lesion level | Within 60 days following 18F-Thretide PET/CT
  The difference in detection rate of 18F-Thretide PET/CT at the lesion level compared with MRI, CT, or bone scanning. Within 60 days following 18F-Thretide PET/CT, either MRI, CT, or bone scan will be performed
sensitivity and specificity | Within 60 days following 18F-Thretide PET/CT
  The sensitivity and specificity of 18F-Thretide PET/CT in the diagnosis of prostate cancer compared with the composite truth standard. Within 60 days following 18F-Thretide PET/CT, either biopsy/surgery, conventional imaging, or locoregional radiation therapy of the 18F-Thretide-suspected lesion(s) will be performed
positive predictive value | Within 60 days following 18F-Thretide PET/CT
  The positive predictive value (PPV) of 18F-Thretide PET/CT in the diagnosis of prostate cancer compared with the composite truth standard. Within 60 days following 18F-Thretide PET/CT, either biopsy/surgery, conventional imaging, or locoregional radiation therapy of the 18F-Thretide-suspected lesion(s) will be performed.
Correct detection rate | Within 60 days following 18F-Thretide PET/CT
  The correct detection rate (CDR) of 18F-Thretide PET/CT imaging in the diagnosis of prostate cancer compared with the composite truth standard. Within 60 days following 18F-Thretide PET/CT, either biopsy/surgery, conventional imaging, or locoregional radiation therapy of the 18F-Thretide-suspected lesion(s) will be performed
Safety evaluation | Within 7 days following 18F-Thretide PET/CT
  The safety will be assessed by the number and percentage of patients with adverse events; Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No